CLINICAL TRIAL: NCT05996666
Title: Early Detection of Primary Liver Cancer Based on cfDNA Methylation: A Multi-Center Case-Control Study (PRIMe-liver)
Brief Title: Primary Liver Cancer Early Detection
Acronym: PRIMe-liver
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Guoyue Lv, Professor of Gastroenterology & Hepatology, The First Hospital of Jilin University
Other Study IDs: RSCD2022015P
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Liver Cancer
Keywords: Early detection; Liver cancer; cell-free DNA (cfDNA); qPCR
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Liver cancer arm: Participants with new diagnosis of liver cancer, from whom blood samples will be collected.
  Interventions: Device: Liver-cancer early detection test
- Benign diseases arm: Participants with benign diseases of cancer, from whom blood samples will be collected.
  Interventions: Device: Liver-cancer early detection test
- Healthy arm: Participants without known presence of malignancies or benign diseases of liver, from whom blood samples will be collected.
  Interventions: Device: Liver-cancer early detection test
- Interfering cancer arm: Participants with new diagnosis of interfering cancer types, from whom blood samples will be collected.
  Interventions: Device: Liver-cancer early detection test

INTERVENTIONS:
Device: Liver-cancer early detection test — Blood collection and liver-cancer early detection test

SUMMARY:
In the recently published multi-center, prospective, single-blind study (THUNDER study), using the methylation signal in cfDNA isolated from the peripheral blood to detect the six types of cancer, the sensitivity for liver cancer detection achieved 87.8%, with a specificity of 98.9%. In this study, a multicenter, case-control study is designed to establish an early cancer detection model based on cfDNA methylation biomarkers using qPCR to detect primary liver cancer and further validate the performance of the model.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all participants

* Individuals aged 18-74 years old
* Individuals capable of giving signed and legally effective informed consent voluntarily

Inclusion Criteria for liver cancer participants:

* Individuals newly diagnosed with or suspected of having liver cancer (including hepatocellular carcinoma [HCC], intrahepatic cholangiocarcinoma [ICC], and combined hepatocellular-cholangiocarcinoma [cHCC-CCA]).
* Individuals without any anti-cancer therapy prior to blood sample collection.

Inclusion Criteria for participants with benign liver diseases:

* Individuals newly diagnosed as benign liver diseases before blood sample collection
* Individuals without curative treatment for the disease before blood sample collection

Inclusion Criteria for participants with interfering cancers:

* Individuals diagnosed with or suspected of having interfering cancer
* Individuals without any anti-cancer therapy prior to blood sample collection

Inclusion Criteria for healthy participants:

* No cancer-related or other clinical symptoms 30 days prior to blood sample collection
* No prior history of benign liver diseases

Exclusion Criteria:

Exclusion Criteria for All the Participants:

* Individuals cannot provide blood samples at the study-specified blood collection sites
* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to blood sample collection
* Recipients of anti-infective treatment within 14 days prior to blood sample collection
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer
* Individuals with a history of malignant tumor

Exclusion Criteria for liver cancer participants:

* Known prior or current diagnosis of other types of malignancies or multiple primary cancers
* No confirmed diagnosis of liver cancer after blood sample collection

Exclusion Criteria for participants with benign liver diseases:

* Individuals with a confirmed diagnosis of a malignant tumor or precancerous lesion
* Individuals who cannot be diagnosed as having benign liver diseases after blood sample collection

Exclusion Criteria for participants with interfering cancers:

* Known prior or current diagnosis of other types of malignancies or multiple primary cancers
* No confirmed diagnosis of any type of interfering cancers after blood sample collection

Exclusion Criteria for healthy participants:

* Prior or ongoing treatment of cancers within 3 years prior to blood sample collection
* Clinically significant or uncontrolled comorbidities

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in this study included subjects with primary liver cancers, benign liver diseases, interfering cancers, and healthy individuals.
Sampling Method: Probability Sample
Enrollment: 701 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Performance of liver cancer early detection model based on selected cfDNA methylation markers using qPCR | 2023.07.01-2023.12.30
  Sensitivity and specificity of liver cancer detection model based on selected cfDNA methylation biomarkers using qPCR in subjects with primary liver cancer or benign liver diseases, interfering cancers and healthy individuals

SECONDARY OUTCOMES:
Performance of the liver cancer early detection model in detecting liver cancer at early stage | 2023.07.01-2023.12.30
  Sensitivity of the liver cancer early detection model in patients with small liver cancer lesions or AFP negative
Performance of liver cancer early detection model in detecting liver cancer at different stages and subtypes | 2023.07.01-2023.12.30
  Sensitivity of the liver cancer early detection model in different stages or different pathological subtypes
Performance of liver cancer early detection model to differentiate non-liver cancers | 2023.07.01-2023.12.30
  Specificity of the liver cancer early detection model to differentiate patients with benign liver diseases or different interfering cancer types from liver cancer
Comparison of currently used biomarkers for liver cancer detection | 2023.07.01-2023.12.30
  Comparison of the sensitivity and specificity of the liver cancer early detection model and other biomarkers of liver cancer in detecting early liver cancer

CONTACTS AND LOCATIONS:
Overall Officials: Tian Yang, Principal Investigator — Eastern Hepatobiliary Surgery Hospital; Nanya Wang, Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - Jilin university first hospital, Changchun, Jilin
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality